CLINICAL TRIAL: NCT03183804
Title: A Follow-up Study to Evaluate the Safety for the Patients With ALLO-ASC-DFU Treatment in Phase 2 Clinical Trial of ALLO-ASC-DFU-201
Brief Title: A Follow-up Study to Evaluate the Safety of ALLO-ASC-DFU in ALLO-ASC-DFU-201 Clinical Trial
Status: Completed | Type: Observational
Sponsor: Anterogen Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: ALLO-ASC-DFU-202
Record Dates: First submitted 2017-06-08; First posted 2017-06-12 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ALLO-ASC-DFU: Subjects with ALLO-ASC-DFU treatment in phase 2 clinical trial of ALLO-ASC-DFU-201
  Interventions: Biological: ALLO-ASC-DFU
- Standard therapy: Subjects with Standard therapy in phase 2 clinical trial of ALLO-ASC-DFU-201
  Interventions: Other: Standard therapy

INTERVENTIONS:
Biological: ALLO-ASC-DFU — Application of ALLO-ASC-DFU sheet to diabetic foot ulcer. This study is a follow-up study without intervention.
  Other Names: Allogeneic mesenchymal stem cells
  Groups: ALLO-ASC-DFU
Other: Standard therapy — Standard therapy conducted for patients with diabetic foot ulcer. This study is a follow-up study without intervention.
  Groups: Standard therapy

SUMMARY:
This is an open-label follow up study to evaluate the safety for the subjects with ALLO-ASC-DFU treatment in phase 2 clinical trial (ALLO-ASC-DFU-201) for 23 months.

DETAILED DESCRIPTION:
This is an open-label follow up study to evaluate the safety for the subjects with ALLO-ASC-DFU treatment in phase 2 clinical trial (ALLO-ASC-DFU-201) for 23 months.

ALLO-ASC-DFU is a hydrogel sheet containing allogenic adipose-derived mesenchymal stem cells. Adipose-derived stem cells have anti-inflammatory effect and release growth factors such as vascular endothelial growth factor (VEGF) and hepatocyte growth factor (HGF), which can enhance wound healing and regeneration of new tissue, finally may provide a new option in treating a Diabetic Foot Ulcer.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are treated with ALLO-ASC-DFU sheet in phase 2 clinical trial of ALLO-ASC-DFU-201.
2. Subjects who are able to give written informed consent prior to study start and to comply with the study requirements.

Exclusion Criteria:

1. Subjects who are considered not suitable for the study by the principal investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject is enrolled who are treated with ALLO-ASC-DFU sheet in phase 2 clinical trial of ALLO-ASC-DFU-201.
Sampling Method: Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2015-12-29 (Actual); Primary Completion 2018-08-17 (Actual); Study Completion 2018-10-24 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | up to 24 months
  Evaluation of AE

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Kyu Han, MD. Ph D., Principal Investigator — Korea University Guro Hospital; Ki-Won Young, MD. Ph D., Principal Investigator — Eulji General Hospital; Hyun-suk Suh, MD. Ph D., Principal Investigator — Asan Medical Center; Jin Woo Lee, MD. Ph D., Principal Investigator — Severance Hospital
Locations (4):
- South Korea (4):
  - Eulji General Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan medical center, Seoul
  - Korea University Guro Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided